CLINICAL TRIAL: NCT04220294
Title: Surgical Site Infection Rate After Subcutaneous Continuous Versus Interrupted Sutures During Cesarean Section.
Brief Title: Subcutaneous Continuous Versus Interrupted Sutures During Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0621-19-RMB
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Suture Line Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupted sutures (Active Comparator): Subcutaneous tissue closure by interrupted sutures.
  Interventions: Procedure: Subcutaneous tissue closure
- Continuous sutures (Active Comparator): Subcutaneous tissue closure by continuous sutures.
  Interventions: Procedure: Subcutaneous tissue closure

INTERVENTIONS:
Procedure: Subcutaneous tissue closure — Subcutaneous tissue closure with 2-0 vicryl suture.

SUMMARY:
A comparison of the rate of surgical site infections after cesarean section depending on the type of suture used for subcutaneous closure-continuous versus interrupted.

DETAILED DESCRIPTION:
Patients at term that are candidates for elective cesarean section will receive an explanation regarding the study and sign informed consent. Patients will then be divided randomly to one of 2 treatment groups based on the type of subcutaneous tissue closure:

1. Interrupted sutures.
2. Continuous sutures. Information regarding medical and obstetric history will be collected for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing elective cesarean section.
* Subcutaneous tissue layer>2 centimeter according to ultrasound.

Exclusion Criteria:

* Non-elective CS.
* Fever during the 48 hours prior to surgery.
* Antibiotic treatment during the 48 hours prior to surgery.
* Inability to give informed consent.
* Preterm delivery (< 37 weeks' gestation).
* Fetal death.
* Known fetal anomalies or placental abnormalities.
* Immunosuppressive conditions.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 1238 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Surgical site infection rate. | From admission up to 6 weeks postpartum.
  Surgical site infection rate.

SECONDARY OUTCOMES:
Rate of re-admission due to surgical site infection. | From admission up to 6 weeks postpartum.
  rate of re-admission within 6 weeks postpartum due to surgical site infection.
Rate of postoperative febrile morbidity. | From admission up to 6 weeks postpartum.
  Rate of maternal body temperature > 38°C.
Rate of maternal fever. | From admission up to 6 weeks postpartum.
  Rate of maternal fever in degrees celsius.
Duration of maternal fever. | From admission up to 6 weeks postpartum.
  Duration of maternal fever in days.
Rate of antibiotic use for the treatment of surgical site infection. | From admission up to 6 weeks postpartum.
  Rate of antibiotic use for the treatment of surgical site infection.
Cesraean section-to-surgical site infection time interval. | From admission up to 6 weeks postpartum.
  Cesraean section-to-surgical site infection time interval in days.
Rate of bacteremia. | From admission up to 6 weeks postpartum.
  Rate of bacteremia.
Rate of sepsis. | From admission up to 6 weeks postpartum.
  Rate of sepsis.
Post-operative duration of hospitalization. | From admission up to 6 weeks postpartum.
  Post-operative duration of hospitalization in days.
Postoperative pain. | From admission up to 6 weeks postpartum.
  Postoperative pain based on the visual analogue scale score ranging from 0-10.
Rate of postoperative anemia. | From admission up to 6 weeks postpartum.
  Rate of a hemoglobin level of under 10 gr/dL
Blood transfusion rates. | From admission up to 6 weeks postpartum.
  Blood transfusion rates (recommended to patients with a postpartum hemoglobin level of under 7 gr/dL or between 7-8 gr/dL if anemia related symptoms are present)
Breastfeeding rates. | From admission up to 6 weeks postpartum.
  Breastfeeding rates.
rate of voiding problems. | From admission up to 6 weeks postpartum.
  Rate of need for either intermittent catheterization or 24-hour foley insertion to void
Venous thromboembolism rates. | From admission up to 6 weeks postpartum.
  Venous thromboembolism rates.
Rate of admission to intensive care unit. | From admission up to 6 weeks postpartum.
  Rates of admission to intensive care unit
Maternal death rate | From admission up to 6 weeks postpartum.
  Maternal death rate.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- Rambam healthcare campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No